CLINICAL TRIAL: NCT02891681
Title: Ultrasound and Near Infrared Imaging for Predicting and Monitoring Neoadjuvant Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 201608101; 7R01EB002136-12 (NIH)
Record Dates: First submitted 2016-08-31; First posted 2016-09-07 (Estimated); Results first posted 2021-02-16 (Actual); Last update posted 2021-02-16 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer; Breast Tumors; Cancer of Breast; Cancer of the Breast; Malignant Neoplasm of Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- NIR/US (Neoadjuvant Chemotherapy Cohort) (Experimental): Patients will have the NIR/US baseline scan performed before their first treatment. The desirable schedule will be >= 7 days after initial biopsy to avoid confounding effects from the biopsy related acute inflammatory response.
  * In addition, patients will also have NIR/US performed at end of cycle 1, end of cycle 2, end of cycle 3, end of cycle 5 (only if treatment regimen changed), and prior to surgery.
  * The number of NIR/US study visits may vary (5-6) depending on the patient's treatment regimen
  Interventions: Device: Optical Tomography Using Near Infrared Diffused Light Assisted with Ultrasound
- NIR/US (Neoadjuvant Endocrine Cohort) (Experimental): Patients will have the NIR/US baseline scan performed before their first treatment. The desirable schedule will be >= 7 days after initial biopsy to avoid confounding effects from the biopsy related acute inflammatory response.
  * In addition, patients will also have NIR/US performed at end of cycle 1, end of cycle 2, end of cycle 3, at time of treatment regimen change (only intended for those who have had a change in their regimen), and prior to surgery.
  * The number of NIR/US study visits may vary (5-6) depending on the patient's treatment regimen
  Interventions: Device: Optical Tomography Using Near Infrared Diffused Light Assisted with Ultrasound

INTERVENTIONS:
Device: Optical Tomography Using Near Infrared Diffused Light Assisted with Ultrasound
  Other Names: NIR/US

SUMMARY:
To determine the accuracy of NIR/US assessment of tumor vasculature and oxygen changes in predicting and monitoring early neoadjuvant treatment response compared to pathological response.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to receive neoadjuvant chemotherapy for the treatment of newly diagnosed, locally advanced breast cancer or scheduled to receive neoadjuvant endocrine therapy with the eventual goal of surgery of newly diagnosed clinical stage II-III ER+ HER2- breast cancer (for the endocrine therapy cohort)
* At least 18 years of age
* Female
* Able to understand and willing to sign an IRB-approved written informed consent document

Exclusion Criteria:

* Pregnant and/or breastfeeding
* Prior history of breast cancer
* Prior history of chest wall radiation
* Prior history of breast reconstruction, reduction, or augmentation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2020-01-23 (Actual); Study Completion 2020-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Quing Zhu, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhu Q, Ademuyiwa FO, Young C, Appleton C, Covington MF, Ma C, Sanati S, Hagemann IS, Mostafa A, Uddin KMS, Grigsby I, Frith AE, Hernandez-Aya LF, Poplack SS. Early Assessment Window for Predicting Breast Cancer Neoadjuvant Therapy using Biomarkers, Ultrasound, and Diffuse Optical Tomography. Breast Cancer Res Treat. 2021 Aug;188(3):615-630. doi: 10.1007/s10549-021-06239-y. Epub 2021 May 10. PMID 33970392
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: An additional arm (NIR/US - Crossover from Endocrine Cohort to Chemotherapy Cohort) was added for results reporting as one participant transitioned from the Endocrine Cohort to the Chemotherapy Cohort because the participant's therapy was changed mid-treatment from Endocrine to Chemotherapy.
Groups:
- NIR/US (Crossover From Endocrine Cohort to Chemotherapy Cohort): Patients will have the NIR/US baseline scan performed before their first treatment. The desirable schedule will be >= 7 days after initial biopsy to avoid confounding effects from the biopsy related acute inflammatory response.
  * In addition, patients will also have NIR/US performed at end of cycle 1, end of cycle 2, end of cycle 3, at time of treatment regimen change (only intended for those who have had a change in their regimen), and prior to surgery.
  * The number of NIR/US study visits may vary (5-6) depending on the patient's treatment regimen
Period: Overall Study
Arm/Group | NIR/US (Neoadjuvant Chemotherapy Cohort) | NIR/US (Neoadjuvant Endocrine Cohort) | NIR/US (Crossover From Endocrine Cohort to Chemotherapy Cohort)
Started | 39 | 1 | 1
Completed | 36 | 1 | 0
Not Completed | 3 | 0 | 1
Not completed — Did not complete all timepoints in Endocrine Cohort | 0 | 0 | 1
Not completed — Developed metastases prior to completing neoadjuvant therapy | 2 | 0 | 0
Not completed — Taken off study after first imaging appointment | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NIR/US (Neoadjuvant Chemotherapy Cohort) | NIR/US (Neoadjuvant Endocrine Cohort) | NIR/US (Crossover From Endocrine Cohort to Chemotherapy Cohort) | Total
Number analyzed (Participants) | 39 | 1 | 1 | 41
Age, Continuous [Median (Full Range); unit: years] | 45 [24 to 73] | 66 [66 to 66] | 53 [53 to 53] | 45 [24 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 1 | 1 | 41
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 38 | 1 | 1 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 1 | 1 | 10
  White | 31 | 0 | 0 | 31
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 39 | 1 | 1 | 41

OUTCOME MEASURES:

1. Primary Outcome: Pathologic Response Based on Miller-Payne Grading System
Description: In the Miller-Payne system, the pathologic response is divided into 5 grades based on comparison of tumor cellularity between pre-neoadjuvant core biopsy and definitive surgical specimen as:
  * grade 1: no change or some alteration to individual malignant cells but no reduction in overall cellularity (pNR)
  * grade 2: a minor loss of tumor cells but overall cellularity still high; up to 30% (pPR)
  * grade 3: between an estimated 30% and 90% reduction in tumor cells (pPR)
  * grade 4: a marked disappearance of tumor cells such that only small clusters or widely dispersed individual cells remain (almost pCR); more than 90% loss of tumor cells
  * grade 5: no malignant cells identifiable in sections from the site of the tumor; only vascular fibroelastonic stroma remains often containing macrophages (pCR) (however, ductal carcinoma in situ (DCIS) may be present)
Time Frame: Up to 6 months
Population: For this outcome measure, the one participant who was in the crossover cohort was counted in the neoadjuvant chemotherapy cohort. Three participants in the neoadjuvant chemotherapy cohort were not evaluable for this outcome measure (2 developed metastases prior to completing neoadjuvant therapy and 1 was taken off study after first imaging appointment).
Measure: Count of Participants; unit: Participants
Arm/Group | NIR/US (Neoadjuvant Chemotherapy Cohort) | NIR/US (Neoadjuvant Endocrine Cohort) | NIR/US (Crossover From Endocrine Cohort to Chemotherapy Cohort)
Number analyzed (Participants) | 37 | 1 | 0
Participants
  Grade 1 | 4 | 1 |
  Grade 2 | 3 | 0 |
  Grade 3 | 8 | 0 |
  Grade 4 | 3 | 0 |
  Grade 5 | 19 | 0 |

ADVERSE EVENTS:
Time Frame: Serious adverse events that occurred within 24 hours of the NIR/US were collected and reported, assessed up to 6 months (~6 months)
Description: Adverse events were not collected for this study. If a serious adverse event was suspected to be caused by the NIR/US scan then it was collected and reported.
Arm/Group | NIR/US (Neoadjuvant Chemotherapy Cohort) | NIR/US (Neoadjuvant Endocrine Cohort) | NIR/US (Crossover From Endocrine Cohort to Chemotherapy Cohort)
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT02891681/Prot_SAP_000.pdf
  • Informed Consent Form (2020-03-25): https://cdn.clinicaltrials.gov/large-docs/81/NCT02891681/ICF_001.pdf